CLINICAL TRIAL: NCT00310024
Title: A Phase I Study of SAHA in Combination With Bortezomib in Relapsed and Refractory Multiple Myeloma
Brief Title: Vorinostat and Bortezomib in Treating Patients With Relapsed or Refractory Multiple Myeloma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02693; GCC 0514; N01CM62204 (NIH); CDR0000466109 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-03-29; First posted 2006-04-03 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Refractory Multiple Myeloma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Vorinostat

ARMS (1):
- Treatment (vorinostat, bortezomib) (Experimental): Patients receive bortezomib IV on days 1, 4, 8, and 11 followed by oral SAHA twice daily on days 4-11. Beginning in course 3, some patients may receive low-dose oral dexamethasone on days 4-8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.
  Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional cohort of 10 patients receive treatment at the MTD.
  Patients undergo blood collection and tumor biopsies periodically during study for pharmacologic and biomarker correlative studies.
  Interventions: Drug: bortezomib; Drug: vorinostat; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Drug: vorinostat — Given orally
  Other Names: L-001079038; SAHA; suberoylanilide hydroxamic acid; Zolinza
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies

SUMMARY:
This phase I trial is studying the side effects and best dose of vorinostat when given together with bortezomib in treating patients with relapsed or refractory multiple myeloma. Vorinostat and bortezomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Giving vorinostat together with bortezomib may kill more cancer cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose (MTD) of vorinostat (SAHA) when given together with bortezomib in patients with relapsed or refractory multiple myeloma (MM).

II. Determine the toxicity of this regimen in these patients.

SECONDARY OBJECTIVES:

I. Determine whether giving SAHA together with bortezomib inhibits histone deacetylation in normal cells (buccal mucosal cells and/or peripheral blood monocytes) as well as in MM cells.

II. Evaluate the effect of dexamethasone when given together with SAHA and bortezomib.

III. Explore molecular mechanisms involved in apoptosis in MM mediated by SAHA and bortezomib.

IV. Correlate change of histone acetylation with clinical outcome in patients treated with this regimen.

OUTLINE: This is a multicenter, dose escalation study of vorinostat (SAHA).

Patients receive bortezomib IV on days 1, 4, 8, and 11 followed by oral SAHA twice daily on days 4-11. Beginning in course 3, some patients may receive low-dose oral dexamethasone on days 4-8. Treatment repeats every 21 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of SAHA until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. An additional cohort of 10 patients receive treatment at the MTD.

Patients undergo blood collection and tumor biopsies periodically during study for pharmacologic and biomarker correlative studies.

After completion of study treatment, patients are followed at least once a month.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and clinically confirmed multiple myeloma

  * Relapsed or refractory disease after prior chemotherapy or transplantation*
* Measurable disease, defined by quantitative immunoglobulin levels in serum and/or urine and bone marrow plasmacytosis

  * Non-secretory disease allowed provided MRI or positron emission tomography or CT scan can accurately measure at least one plasmacytoma lesion
* No known CNS involvement
* Life expectancy > 3 months
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Absolute neutrophil count ≥ 1,000/mm³ (unless myelosuppression is secondary to bone marrow plasmacytosis [> 80% involvement])
* Platelet count ≥ 50,000/mm³ (unless myelosuppression is secondary to bone marrow plasmacytosis [> 80% involvement])
* Bilirubin ≤ 2 times upper limit of normal (ULN)
* AST and ALT ≤ 2 times ULN
* Creatinine < 2 mg/dL OR creatinine clearance > 40 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Able to swallow pills
* Patients with a history of seizures are eligible provided seizures are under adequate control with non-enzyme inducing anticonvulsant medication
* No history of allergic reactions attributed to study agents
* No sensory or motor neuropathy ≥ grade II
* No uncontrolled current illness including, but not limited to, the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness or social situation that would limit study compliance
* No grade 3 QT prolongation (i.e., > 500 msec) at baseline
* See Disease Characteristics
* Prior bortezomib allowed
* At least 2 weeks since prior therapy for multiple myeloma
* Concurrent growth factors (filgrastim [G-CSF] and epoetin alfa) to sustain peripheral blood counts (during the first course of therapy only) allowed
* Concurrent steroid therapy (≤ 20 mg of prednisone) for patients requiring chronic use for disorders other than myeloma allowed
* No concurrent combination antiretroviral therapy for HIV-positive patients
* No other concurrent investigational or commercial agents or therapies for this malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2005-11; Primary Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of SAHA in combination with bortezomib determined by dose-limiting toxicities | 21 days

SECONDARY OUTCOMES:
Inhibition of histone deacetylation | Up to 1 month
Response | Up to 1 month
  The estimates and the corresponding 90% confidence intervals will be calculated.
Survival (disease specific and overall) | Up to 1 month
  Will be estimated using the Kaplan-Meir method.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Badros, Principal Investigator — University of Maryland Greenebaum Cancer Center
Locations (1):
- University of Maryland Greenebaum Cancer Center, Baltimore, Maryland, United States